CLINICAL TRIAL: NCT07303166
Title: Qualitative Study Exploring the Determinants Involved in the Management of Osteoporosis in Frail Elderly People by Doctors in Alsace Who Had Access to a Practical Guide on Osteoporosis
Brief Title: Qualitative Study Exploring the Determinants Involved in the Management of Osteoporosis in Frail Elderly People
Acronym: QualiFichOs
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 9482
Record Dates: First submitted 2025-12-11; First posted 2025-12-24 (Actual); Last update posted 2025-12-24 (Actual); Status verified 2025-12

CONDITIONS: Osteoporosis
Keywords: Osteoporosis; Osteoporosis in elderly people
MeSH Terms: conditions — Osteoporosis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The aging population is associated with an increase in the number of elderly people as well as in chronic diseases, particularly osteoporosis and its fracture consequences, which lead to a decline in quality of life and life expectancy. Improved management of osteoporosis would help reduce the morbidity and mortality associated with this disease.

ELIGIBILITY:
Inclusion Criteria:

* Alsatian doctors treating elderly patients with osteoporosis
* Who have had the opportunity to use the practical guide on osteoporosis

Exclusion Criteria:

- A doctor who has never had the opportunity to use the practical guide on osteoporosis.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Alsatian doctors treating elderly patients with osteoporosis
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-11-15 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-02 (Estimated)

PRIMARY OUTCOMES:
Identify the factors promoting and hindering the use of a practical guide on the management of osteoporosis | Up to 12 months
  Identify the factors promoting and hindering the use of a practical guide on the management of osteoporosis

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Gériatrie Aiguë - CHU de Strasbourg - France, Strasbourg, France